CLINICAL TRIAL: NCT03605342
Title: Optimal Treatment of Veterans With PTSD and Comorbid Opiate Use Disorder (OUD)
Brief Title: Optimal Treatment of Veterans With PTSD and Comorbid OUD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBB-010-17F
Record Dates: First submitted 2018-06-29; First posted 2018-07-30 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Post-Traumatic Stress Disorders; Opiate Use Disorder
Keywords: PTSD; Opiate Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Buprenorphine

STUDY DESIGN:
Intervention Model Description: This study is a 14-week, open-label randomization: 1) buprenorphine (BUP) + CPT-C vs (2) BUP + IDC. Phase I: buprenorphine induction and stabilization for all participants. Participants starting dose 2mg/0.5 mg BUP/NLX this will increase as needed up to 24 mg per day. Phase II: randomization to CPT vs. IDC (x12 weeks). Phase III: Subjects will be referred to one of the buprenorphine clinics and will be referred for ongoing treatment for PTSD if they choose, including the option for CPT-C for those who did not receive this during the study. Participants will be seen on a daily basis (excluding weekends) for the initial 5-7 day induction. Once subjects are on maintenance dose of BUP/NLX, they will be seen weekly by study Registered Nurse (RN) for the first 4 weeks, biweekly for a month then monthly for symptom evaluation, and medication refill.
Who Masked: Outcomes Assessor
Masking Description: To fully assess and appreciate complex symptomatology in this patient population, assessments were selected to have both relevance to the investigators' study of PTSD and comorbid OUD. Assessments will be done by an Independent Evaluator (IE) blind to treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buprenorphine + CPT-C (Active Comparator): Buprenorphine induction and stabilization for all participants (x1 week). Participants will be started at a dose of 2mg/0.5 mg BUP/NLX and this dose will be increased as needed for stabilization of opioid withdrawal symptoms up to 24 mg per day, then CPT-C for 12 weeks.
  Interventions: Drug: Buprenorphine; Behavioral: Cognitive Processing Therapy (CPT)
- Buprenorphine + IDC (Active Comparator): Buprenorphine induction and stabilization for all participants (x1 week). Participants will be started at a dose of 2mg/0.5 mg BUP/NLX and this dose will be increased as needed for stabilization of opioid withdrawal symptoms up to 24 mg per day, then IDC for 12 weeks
  Interventions: Drug: Buprenorphine; Behavioral: Individual Drug Counseling (IDC)

INTERVENTIONS:
Drug: Buprenorphine — Participants will be started at a dose of 2mg/0.5 mg BUP/NLX and this dose will be increased as needed for stabilization of opioid withdrawal symptoms up to 24 mg per day, which is standard practice.
Behavioral: Cognitive Processing Therapy (CPT) — CPT-C is a manualized, 12-session 1:1 cognitive therapy that has been designed for patients with PTSD. In this study the sessions will be conducted weekly. CPT-C uses Socratic questioning targeting distorted cognitions such as self-blame, hindsight bias, and other guilt cognitions. CPT-C is focused on the cognitive components of the therapy without exposure.
  Arms: Buprenorphine + CPT-C
Behavioral: Individual Drug Counseling (IDC) — IDC will serve as the control group. The current standard of treatment for Veterans entering buprenorphine maintenance is to do drug counseling. Standard counseling is the primary means to achieve goals. IDC uses a semi-structured, time-limited addictions-counseling model in a 1:1 setting. The IDC manual provides an organized, concise version of what is currently practiced by most addiction counselors.
  Arms: Buprenorphine + IDC

SUMMARY:
The objective of this study is to test a standard psychotherapy for PTSD in Veterans who also suffer from Opiate Use Disorder (OUD). Specifically, this study will test whether Cognitive Processing Therapy (CPT)-C is more effective in treating PTSD, compared to a control group (Individual Drug Counseling (IDC); which approximates treatment as usual), among Veterans with PTSD and comorbid OUD who are maintained on buprenorphine.

The study has three phases. In Phase I: induction to buprenorphine/naloxone (BUP/NLX) maintenance. Phase II: treatment. During this phase participants will be randomly assigned to CPT-C or IDC for 12 weeks. They will be seen weekly for psychotherapy and also regularly (weekly, then biweekly, then monthly) for buprenorphine management, symptom evaluation, and medication refill. After completing treatment participants will be referred to a buprenorphine clinic for ongoing care. Phase III: follow-up.

Approximately 160 male and female Veterans (18-65 years old) with PTSD and comorbid opiate use disorder (OUD) will be enrolled in this study. Recruitment will be through VA clinics, word-of-mouth, referrals from area programs and by advertisement. Veterans who are interested will complete a brief pre-screening and detailed in-person screening. After completing the screening process, all eligible participants will be started on buprenorphine maintenance and once withdrawal symptoms are stabilized, participants will be randomly assigned to 1 of 2 conditions (CPT-C or IDC) for 12 weeks. Veterans who are already on BUP/NLX will be allowed to participate and will start at Phase II of the study, after completing the screening.

DETAILED DESCRIPTION:
The purpose of this study is to test whether Cognitive Processing Therapy (CPT-C) is more effective than Individual Drug Counseling (IDC), which is standard counseling, for the treatment of PTSD among Veterans with PTSD and comorbid opioid use disorder who are also maintained on buprenorphine. The investigators propose to conduct a randomized, controlled trial and Veterans (n=160) diagnosed with PTSD and comorbid OUD will be randomized to one of 2 groups: (a) buprenorphine and CPT-C or (b) buprenorphine and IDC (treatment as usual).

Primary Aim 1:.To test whether CPT-C is more effective than IDC in treating symptoms of PTSD among Veterans with OUD maintained on buprenorphine. PTSD symptoms will be measured using the PTSD Checklist - Military version (PCL-5) and confirmed by the Clinician Administered PTSD Scale using the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria (CAPS-5).

Secondary Aim 1: To test whether CPT-C is more effective than IDC in reducing opioid use among Veterans with PTSD and comorbid OUD maintained on buprenorphine. Opioid use will be measured using the Timeline Follow-back (TLFB) and confirmed by urine toxicology results.

Exploratory Aims: To examine if treatment groups differ in 1) retention, measured by days in treatment, 2) psychosocial functioning, measured by the Veterans RAND 12-Item Short Form Health Survey (VR-12), 3) sleep as measured by the Insomnia Severity Index (ISI), since sleep disturbance is a hallmark of PTSD and during early abstinence from opioids, and 4) Because of the high comorbidity between PTSD and chronic pain the investigators will explore this relationship and will measure pain intensity (measured by the Numeric Rating Scale (NRS), and functional impairment using the Patient-Reported Outcomes Measurement Information System (PROMIS-29) longitudinally over the course of treatment. Follow up will be conducted 1 and 3 months after completion of the study to evaluate durability of effect on PTSD symptoms (measured as changes in PTSD symptoms), opioid use and treatment utilization.

This study will be a randomized, open-label clinical trial. The study has three phases. In Phase I: induction to buprenorphine/naloxone (BUP/NLX) maintenance. Phase II: treatment. During this phase participants will be randomly assigned to CPT-C or IDC for 12 weeks. They will be seen weekly for psychotherapy and also regularly (weekly, then biweekly, then monthly) for buprenorphine management, symptom evaluation, and medication refill. After completing treatment participants will be referred to a buprenorphine clinic for ongoing care. Phase III: follow-up.

Approximately 160 male and female Veterans (18-65 years old) with PTSD and comorbid opiate use disorder (OUD) will be enrolled in this study. Recruitment will be through VA clinics, word-of-mouth, referrals from area programs and by advertisement. Veterans who are interested will complete a brief pre-screening and detailed in-person screening (including: consent, lab work, interview with clinician including the Structured Clinical Interview for DSM-5 (SCID-5) and Clinician Administered PTSD Scale for DSM-5 (CAPS-5), medical and psychiatric history). After completing the screening process, all eligible participants will be started on buprenorphine maintenance and once withdrawal symptoms are stabilized, participants will be randomly assigned to 1 of 2 conditions (CPT-C or IDC) for 12 weeks. Veterans who are already on BUP/NLX will be allowed to participate and will start at Phase II of the study, after completing the screening. The investigators will use mixed effects models to assess changes in PTSD symptoms and opiate use over time. Treatments will be used as between-subject factors and time (in weeks) will be used as a within-subject factor. The primary outcome variables will be PTSD symptoms as measured by the PCL-5 and CAPS scales. The secondary outcome variables will be frequency of opiate use generated from the TLFB and confirmed with urine toxicology results at each medication visit (weeks 1-4, 6,8, 12) and follow-up.

Potential benefits of participation in this study may include a reduction in PTSD symptoms. However, there is no guarantee or promise that participants will receive any benefit from participation in this study.

Since 11 September 2001, more than 1.5 million Service Members have deployed more than 2 million times in support of combat operations in Afghanistan and Iraq. One of the signature injuries from these operations is PTSD. Various reports of the post-deployment health-related needs estimated that 20% of Veterans returning from deployment will have symptoms of PTSD or related behavioral health conditions. In addition, the prescription opioid epidemic has seriously affected Veterans, and Veterans with PTSD are more likely to abuse opioids and to have high-risk behaviors. Nevertheless, treating comorbid PTSD and OUD has not been systematically tested. This study proposes to test an evidence based psychotherapy for PTSD vs. individual drug counseling in Veterans given opioid maintenance treatment who have both PTSD and OUD.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of PTSD as determined by an independent evaluator assessment using CAPS-5.
* Opioid Use Disorder diagnosed by Structured Clinical Interview for DSM-5 (SCID-V)

  * To meet entry criteria for buprenorphine treatment:

    * will also have documented prior treatment for opioid use disorder
    * history of opioid withdrawal or signs of opiate withdrawal as evidenced by a Clinical Opiate Withdrawal Scale (COWS) score of 7 or greater
    * a positive urine toxicology for opioids
* Medically and neurologically healthy on the basis of:

  * history
  * physical examination
  * EKG
  * screening blood tests (CBC w/ differential, Thyroid-stimulating hormone (TSH), Free-T4, aspartate aminotransferase (AST), alanine aminotransferase (ALAT), Gamma-glutamyl transferase (GGT), blood urea nitrogen (BUN), creatinine, calcium, phosphorous, magnesium, total protein, albumin, electrolytes, urinalysis, urine toxicology, beta-HCG)
* For women, negative pregnancy test and use of acceptable method of contraception

Exclusion Criteria:

* Females who are pregnant or lactating
* Veterans with a current unstable medical condition such as:

  * neurological
  * cardiovascular
  * endocrine
  * renal
  * liver
  * or thyroid pathology (e.g. abnormal BUN and creatinine, and unmanaged hypertension with BP > 200/120) which in the opinion of the physician would preclude the patient from fully cooperating or be of potential harm during the course of the study
* Veterans who meet current criteria for the following diagnoses (bipolar disorders, schizophrenia and schizophrenia spectrum and psychotic disorders) as determined by the SCID-V
* Veterans who have significant current suicidal or homicidal risks necessitating a higher level of care
* Those with known allergy or intolerance to buprenorphine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismene L. Petrakis, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Petrakis IL, Meshberg-Cohen S, Nich C, Kelly MM, Claudio T, Jane JS, Pisani E, Ralevski E. Cognitive processing therapy (CPT) versus individual drug counseling (IDC) for PTSD for veterans with opioid use disorder maintained on buprenorphine. Am J Addict. 2024 Sep;33(5):525-533. doi: 10.1111/ajad.13557. Epub 2024 Apr 16. PMID 38624259

RESULTS

PARTICIPANT FLOW:
Groups:
- Buprenorphine + CPT-C: Buprenorphine (BUP) induction and stabilization for all participants (x1 week). Participants will be started at a dose of 2mg/0.5 mg buprenorphine and naloxone (BUP/NLX) and this dose will be increased as needed for stabilization of opioid withdrawal symptoms up to 24 mg per day, then CPT-C for 12 weeks.
  Buprenorphine: Participants will be started at a dose of 2mg/0.5 mg BUP/NLX and this dose will be increased as needed for stabilization of opioid withdrawal symptoms up to 24 mg per day, which is standard practice.
  Cognitive Processing Therapy (CPT): CPT-C is a manualized, 12-session 1:1 cognitive therapy that has been designed for patients with PTSD. In this study the sessions will be conducted weekly. CPT-C uses Socratic questioning targeting distorted cognitions such as self-blame, hindsight bias, and other guilt cognitions. CPT-C is focused on the cognitive components of the therapy without exposure.
- Buprenorphine + IDC: Buprenorphine (BUP) induction and stabilization for all participants (x1 week). Participants will be started at a dose of 2mg/0.5 mg buprenorphine and naloxone (BUP/NLX) and this dose will be increased as needed for stabilization of opioid withdrawal symptoms up to 24 mg per day, then IDC for 12 weeks
  Buprenorphine: Participants will be started at a dose of 2mg/0.5 mg BUP/NLX and this dose will be increased as needed for stabilization of opioid withdrawal symptoms up to 24 mg per day, which is standard practice.
  Individual Drug Counseling (IDC): IDC will serve as the control group. The current standard of treatment for Veterans entering buprenorphine maintenance is to do drug counseling. Standard counseling is the primary means to achieve goals. IDC uses a semi-structured, time-limited addictions-counseling model in a 1:1 setting. The IDC manual provides an organized, concise version of what is currently practiced by most addiction counselors.
Period: Overall Study
Arm/Group | Buprenorphine + CPT-C | Buprenorphine + IDC
Started | 20 | 18
Completed | 10 | 10
Not Completed | 10 | 8
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine + CPT-C | Buprenorphine + IDC | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (12.74) | 48.44 (11) | 46.89 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 20 | 15 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 15 | 13 | 28
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 18 | 38
Trauma Types [Count of Participants; unit: Participants]
  Combat Exposure | 10 | 6 | 16
  Sexual Assault | 5 | 5 | 10
  Serious Accident/Assault | 3 | 4 | 7
  Witnessing Severe Injury or Death | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS-5)
Description: Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (CAPS-5) is a structured diagnostic interview. The scale also assesses social and occupational functioning, dissociation symptoms, and the validity of symptom reports. The CAPS-5 uses a single 5-point ordinal rating scale to measure symptom severity. Symptom severity ratings combine information about symptom frequency and intensity obtained by the interviewer. The CAPS-5 requires approximately 40 minutes to administer.
  Scores can range from 0 (minimum score) - 80 (maximum score) with higher scores indicating greater severity. (0-19=Asymptomatic/few symptoms very mild PTSD, 20-39=Sub-threshold/mild PTSD, 40-59=Threshold PTSD/moderate PTSD, 60-79=Severe PTSD, 80=Extreme PTSD)
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Buprenorphine + CPT-C | Buprenorphine + IDC
Number analyzed (Participants) | 20 | 18
units on a scale | 31.95 (2.62) | 34.38 (2.76)

2. Primary Outcome: PTSD Checklist - Military Version (PCL-5) Total Score
Description: PCL-5 will be used to collect information on PTSD symptoms. The PCL-5 is a 20-item self-report measure, selected for its dimensional sensitivity, with higher scores reflecting greater PTSD severity. Scoring is based on how much the patient has been bothered by the symptoms on a scale from "0 = not at all" to "4 = extremely." Items are summed to provide a total severity score (range 0-80). PCL-5 score between 31-33 is indicative of PTSD.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Buprenorphine + CPT-C | Buprenorphine + IDC
Number analyzed (Participants) | 20 | 18
units on a scale | 44.80 (3.66) | 45.44 (3.86)

3. Primary Outcome: Clinician Administered PTSD Scale (CAPS-5)
Description: as for outcome 1
Time Frame: Week 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Buprenorphine + CPT-C | Buprenorphine + IDC
Number analyzed (Participants) | 20 | 18
units on a scale | 29.59 (3.64) | 27.12 (3.25)

4. Primary Outcome: PTSD Checklist - Military Version (PCL-5) Total Score
Description: as for outcome 2
Time Frame: Week 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Buprenorphine + CPT-C | Buprenorphine + IDC
Number analyzed (Participants) | 20 | 18
units on a scale | 34.17 (4.23) | 29.39 (4.30)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Events are not listed separately for each intervention but are reported by trial arm.
Arm/Group | Buprenorphine + CPT-C | Buprenorphine + IDC
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT03605342/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT03605342/ICF_001.pdf